CLINICAL TRIAL: NCT02064556
Title: A Randomized, Open-label, Multiple Doses, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction and Safety of Amlodipine Between Free Combination of Amlodipine and Candesartan and Amlodipine Monotherapy in Healthy Male Volunteers
Brief Title: CKD-330 Drug-Drug Interaction Study (Amlodipine)
Acronym: CKD-330(A)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 144HPS13012
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A(Amlodipine 10mg) (Experimental): Amlodipine 10mg 1T, PO, QD for 9days
  Interventions: Drug: Amlodipine 10mg/Candesartan 32mg
- B(Amlodipine 10mg/Candesartan 32mg) (Experimental): Amlodipine 10mg 1T, PO, QD for 9days/Candesartan 32mg 1T, PO, QD for 9days
  Interventions: Drug: Amlodipine 10mg

INTERVENTIONS:
Drug: Amlodipine 10mg — Amlodipine 10mg 1T, PO, QD for 9days
  Other Names: Norvasc Tab. 10mg
  Arms: B(Amlodipine 10mg/Candesartan 32mg)
Drug: Amlodipine 10mg/Candesartan 32mg — Amlodipine 10mg 1T, PO, QD for 9days/Candesartan 32mg 1T, PO, QD for 9days
  Other Names: Norvasc Tab. 10mg/Atacand Tab. 32mg
  Arms: A(Amlodipine 10mg)

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction and safety of Amlodipine between free combination of Amlodipine and Candesartan and Amlodipine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer is between 20 and 45 years of age(inclusive) at the pre-study(screening).
2. Volunteer who has 19kg/m² ≤ BMI(Body Mass Index) ≤ 26kg/m²
3. When volunteer in screening, Must include under the items.

   1. 100 mmHg ≤ sitting SBP <140 mmHg
   2. 60 mmHg ≤ sitting DBP < 90 mmHg
   3. 45 bpm ≤ Pulse < 95 bpm
4. Those who decided to join the clinical trials by themselves and to comply with the precautions written consent.

Exclusion Criteria:

1. A previous history or present of clinically significant liver, renal, gastro-intestinal, pulmonary, musculoskeletal, endocrine, neuropsychiatric, hemato-oncological, cardiovascular disease.
2. Have a gastrointestinal disease history that can affect drug absorption(Crohn's disease, Ulcers, GERD, Gastritis, etc.) or surgery (except simple appendectomy or hernia surgery).
3. The history of clinically significant hypersensitivity reaction about Investigational drugs and foods.
4. The history of drug abuse or drug abuse showed a positive for urine drug test.
5. Taking drugs have received any other investigational drug within 90 days prior to the first dosing and metabolizing enzyme inducers or inhibitors such as barbitals within 30 days prior to the first dosing.
6. Whole blood donation within 60 days prior to the first dosing or plasma donation within 30 days prior to the first dosing.
7. Taking drugs that clinical trials expected to affect within 14days or taking food containing caffeine, grapefruit within 7days before the first dosing.
8. A heavy alcohol consumer(alcohol>3cup/day or 3times/week within last 1month)
9. A heavy smoker(cigarette>10cigarettes/day)
10. The subject has positive results of serum tests(Hepatitis B, C, HIV Test, Syphilis).
11. Have the Liver enzyme levels(AST, ALT) or Bilirubin, total results greater than 1.5 times the UNL.
12. Have the result of Creatinine clearance is less than 80mL/min(Cockcroft-Gault equation applicable).
13. The result of 12-lead ECG in screening test is QTc>450msec.
14. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of Amlodipine | 1D 0h, 8D 0h, 9D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h, 10D 0h, 11D 0h
Cmax,ss of Amlodipine | 1D 0h, 8D 0h, 9D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h, 10D 0h, 11D 0h

SECONDARY OUTCOMES:
Tmax,ss of Amlodipine | 1D 0h, 8D 0h, 9D 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h, 10D 0h, 11D 0h

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea